CLINICAL TRIAL: NCT03056612
Title: Predicting Acute-on-Chronic Liver Failure in Cirrhosis (PREDICT) Study
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Jonel Trebicka (Other)
Responsible Party: Sponsor-Investigator, Jonel Trebicka, Principal Investigator EFCLIF, European Foundation for Study of Chronic Liver Failure
Organization: European Foundation for Study of Chronic Liver Failure (Other)
Other Study IDs: PREDICT
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Liver Cirrhosis With Acute Decompensation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral serum, plasma, PBMC/PMN, urine, hair (in case of alcohol abuse), ascites (if any), stool, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 patients with high risk of ACLF development (CLIF-C AD score ≥ 50)
  Interventions: Other: Observation protocol
- Group 2: Group 2 patients with low risk of ACLF (CLIF-C AD score <50)
  Interventions: Other: Observation protocol
- ACLF: ACLF-patients were specified the patients who were admitted at hospital with ACLF,
  Interventions: Other: Observation protocol

INTERVENTIONS:
Other: Observation protocol — The whole cohort will be followed for 3 months, while Group 1 will be followed more closely.

SUMMARY:
The aim of this study is to assess prospectively the critical period prior to the development of Acute-on-Chronic Liver Failure (ACLF) (1), to uncover mechanistic and pathophysiological processes associated with the development and clinical course of ACLF (2) and to identify the precipitating events of ACLF (3).

DETAILED DESCRIPTION:
1. This International-European, investigator-initiated, multicenter, prospective, observational study will be performed in centers that belong to the European Foundation for the Study of Chronic Liver failure (EF-CLIF)-European Association for Study of the Liver (EASL)-EASL-CLIF Consortium.
2. The population of patients would include ca. 1,200 cirrhotic patients over a twelve-months period. These patients will be admitted/referred to the study center because of acute decompensation (AD) of cirrhosis (ascites, overt encephalopathy, GI-hemorrhage, new onset of non-obstructive jaundice and/or bacterial infections), without ACLF (as defined according to the Canonic study ) at hospitalization.
3. After the enrolment visit, the patients will be stratified into two groups: Group 1 patients with high risk of ACLF development (CLIF-C AD score ≥ 50) and in Group 2 patients with low risk of ACLF (CLIF-C AD score <50). The whole cohort will be followed for 3 months, while Group 1 will be followed more closely. Development of ACLF is an end-point and in this case a final visit 7-10 days after ACLF development is planned. Data on liver transplantation, mortality and causes of mortality 3 months, 6 months and 12 months will be collected in the whole cohort.
4. Prospective collection of biological material and performance of ancillary studies investigating predictors for development and pathogenesis of ACLF.

Specific goals of the study:

* To identify early clinical predictors, biomarkers, mechanisms and precipitating events during the critical period prior to and involved in the development and clinical course of ACLF (with special emphasis to medical trajectory and drug history) in patients admitted/referred to study center with acute decompensation of cirrhosis (ascites, GI-hemorrhage, overt encephalopathy, new onset of non-obstructive jaundice and/or bacterial infections) and the chronological relationship of the events with occurrence and dynamics of ACLF development.
* To develop a score predicting ACLF development (CLIF-PREDICT score) and assess 28-day, 90-day, 6-month and 1-year all-cause mortality in cirrhotic patients with acute AD, but without ACLF.
* To serve as a core (hub) study for prospective ancillary studies regarding diagnosis, prognosis and pathogenesis of AD and ACLF.

Main endpoints

* Assessment of the critical period prior to ACLF development

  * Characterization of mechanisms responsible for ACLF development
  * Predictors of clinical course dynamics of ACLF evolution and mortality.
  * Identification and role of precipitating events for ACLF development.
* To elaborate a CLIF-PREDICT score 2. Secondary endpoints
* Prospective core ancillary studies to investigate the pathogenesis of ACLF.

ELIGIBILITY:
Inclusion Criteria:

The patients admitted/referred to study center with AD of cirrhosis (ascites, overt encephalopathy, new onset of non-obstructive jaundice, GI-hemorrhage and/or bacterial infections), but without ACLF (as defined according to the CANONIC study) at study inclusion.

Exclusion Criteria:

1. Presence of ACLF at inclusion;
2. Pregnancy;
3. Age <18 years;
4. Patients with acute or subacute liver failure without underlying cirrhosis;
5. Patients with cirrhosis who develop decompensation in the postoperative period following partial hepatectomy;
6. Evidence of current malignancy except for non-melanocytic skin cancer and hepatocellular carcinoma within Milan criteria;
7. Presence or history of severe extra-hepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe heart disease (NYHA > II); severe chronic pulmonary disease (GOLD > III), severe neurological and psychiatric disorders);
8. HIV-positive patients
9. Previous liver or other transplantation
10. Admission/referral of more than 72 hours before inclusion
11. Patients who decline to participate or who cannot provide prior written informed consent and when there is documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent;
12. Physician´s denial (e.g. the investigator considers that the patient will not follow the protocol scheduled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of patients would include ca. 1,200 cirrhotic patients over a twelve-months period. These patients will be admitted/referred to the study center because of acute decompensation of cirrhosis (ascites, overt encephalopathy, GI-hemorrhage, new onset of non-obstructive jaundice and/or bacterial infections), without ACLF (as defined according to the CANONIC study ) at hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 1314 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients developing ACLF within 12 weeks and severity of ACLF development | 12 weeks
  * Characterization of mechanisms responsible for ACLF development
  * Predictors of clinical course dynamics of ACLF evolution and mortality.
  * Identification and role of precipitating events for ACLF development.

SECONDARY OUTCOMES:
Score to PREDICT ACLF | 12 weeks
  -Calculate a Score to predict ACLF

CONTACTS AND LOCATIONS:
Locations (45):
- Austria (3):
  - Medical University Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Belgium (4):
  - University Hospital Antwerp, Antwerp
  - C.U.B Erasmo, Brussels
  - Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Hvidovre University Hospital, Copenhagen
- France (3):
  - Hospital Jean Verdier, Bondy
  - Hopital Beaujon, Paris
  - Hopital Paul Brousse, Paris
- Germany (8):
  - RTWH Aachen, Aachen
  - University Hospital Bonn, Bonn
  - JW Goethe University Hospital, Frankfurt am Main
  - University Hospital Halle-Wittenberg, Halle
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - University Hospital Leipzig, Leipzig
  - University Hospital Munich LMU, Munich
- University of Debrecen, Debrecen, Hungary
- Italy (5):
  - University of Bologna, Bologna
  - Internal Medicine PO Ostuni, Brindisi
  - University Clinic Padova, Padua
  - Universita Sapienza, Rome
  - A.O.U. Torino, Torino
- Leiden University Medical Center, Leiden, Netherlands
- CHTMAD Vila Real, Vila Real, Portugal
- Pavol Jozef Sfarik University Kosice/Roosevelt Hospital Bystrica, Košice, Slovakia
- Spain (6):
  - Hospital Clinic y Provencial de Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Virgen del Rocio, Seville
- Switzerland (3):
  - Inselspital, Bern
  - Hôpitaux Universitaires Geneve, Geneva
  - Cantonal Hospital St. Gallen, Sankt Gallen
- Marsara University, Istanbul, Turkey (Türkiye)
- United Kingdom (6):
  - Birmingham University Hospitals, Birmingham
  - Imperial College, London
  - King´s College, London
  - Royal Free Hospital, London
  - Nottingham University Hospitals, Nottingham
  - Derriford Hospital, Plymouth Hospitals Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Espen L, Brol MJ, Close L, Schierwagen R, Gu W, Keller MI, Balogh B, Fullam A, De Coninck L, Nakamura T, Kuhn M, Bork P, Laleman W, Bajaj JS, Papp M, Schnabl B, Trebicka J, Matthijnssens J; MICROB-PREDICT. L actococcus A phages predict ACLF while Enterococcus B phages predict bacterial infection in decompensated cirrhosis. JHEP Rep. 2025 Oct 10;8(1):101622. doi: 10.1016/j.jhepr.2025.101622. eCollection 2026 Jan. PMID 41438339
- [Derived] Weiss E, de la Pena-Ramirez C, Aguilar F, Lozano JJ, Sanchez-Garrido C, Sierra P, Martin PI, Diaz JM, Fenaille F, Castelli FA, Gustot T, Laleman W, Albillos A, Alessandria C, Domenicali M, Caraceni P, Piano S, Saliba F, Zeuzem S, Gerbes AL, Wendon JA, Jansen C, Gu W, Papp M, Mookerjee R, Gambino CG, Jimenez C, Giovo I, Zaccherini G, Merli M, Putignano A, Uschner FE, Berg T, Bruns T, Trautwein C, Zipprich A, Banares R, Presa J, Genesca J, Vargas V, Fernandez J, Bernardi M, Angeli P, Jalan R, Claria J, Junot C, Moreau R, Trebicka J, Arroyo V. Sympathetic nervous activation, mitochondrial dysfunction and outcome in acutely decompensated cirrhosis: the metabolomic prognostic models (CLIF-C MET). Gut. 2023 Aug;72(8):1581-1591. doi: 10.1136/gutjnl-2022-328708. Epub 2023 Feb 14. PMID 36788015
- [Derived] Trebicka J, Fernandez J, Papp M, Caraceni P, Laleman W, Gambino C, Giovo I, Uschner FE, Jansen C, Jimenez C, Mookerjee R, Gustot T, Albillos A, Banares R, Jarcuska P, Steib C, Reiberger T, Acevedo J, Gatti P, Shawcross DL, Zeuzem S, Zipprich A, Piano S, Berg T, Bruns T, Danielsen KV, Coenraad M, Merli M, Stauber R, Zoller H, Ramos JP, Sole C, Soriano G, de Gottardi A, Gronbaek H, Saliba F, Trautwein C, Kani HT, Francque S, Ryder S, Nahon P, Romero-Gomez M, Van Vlierberghe H, Francoz C, Manns M, Garcia-Lopez E, Tufoni M, Amoros A, Pavesi M, Sanchez C, Praktiknjo M, Curto A, Pitarch C, Putignano A, Moreno E, Bernal W, Aguilar F, Claria J, Ponzo P, Vitalis Z, Zaccherini G, Balogh B, Gerbes A, Vargas V, Alessandria C, Bernardi M, Gines P, Moreau R, Angeli P, Jalan R, Arroyo V; PREDICT STUDY group of the EASL-CLIF CONSORTIUM. PREDICT identifies precipitating events associated with the clinical course of acutely decompensated cirrhosis. J Hepatol. 2021 May;74(5):1097-1108. doi: 10.1016/j.jhep.2020.11.019. Epub 2020 Nov 20. PMID 33227350
- [Derived] Trebicka J, Fernandez J, Papp M, Caraceni P, Laleman W, Gambino C, Giovo I, Uschner FE, Jimenez C, Mookerjee R, Gustot T, Albillos A, Banares R, Janicko M, Steib C, Reiberger T, Acevedo J, Gatti P, Bernal W, Zeuzem S, Zipprich A, Piano S, Berg T, Bruns T, Bendtsen F, Coenraad M, Merli M, Stauber R, Zoller H, Ramos JP, Sole C, Soriano G, de Gottardi A, Gronbaek H, Saliba F, Trautwein C, Ozdogan OC, Francque S, Ryder S, Nahon P, Romero-Gomez M, Van Vlierberghe H, Francoz C, Manns M, Garcia E, Tufoni M, Amoros A, Pavesi M, Sanchez C, Curto A, Pitarch C, Putignano A, Moreno E, Shawcross D, Aguilar F, Claria J, Ponzo P, Jansen C, Vitalis Z, Zaccherini G, Balogh B, Vargas V, Montagnese S, Alessandria C, Bernardi M, Gines P, Jalan R, Moreau R, Angeli P, Arroyo V; PREDICT STUDY group of the EASL-CLIF Consortium. The PREDICT study uncovers three clinical courses of acutely decompensated cirrhosis that have distinct pathophysiology. J Hepatol. 2020 Oct;73(4):842-854. doi: 10.1016/j.jhep.2020.06.013. Epub 2020 Jul 13. PMID 32673741